CLINICAL TRIAL: NCT06139562
Title: Two Different Dietary Approaches In Body Composition And Serum Hormone Levels: Time-Restricted And Extended Feeding
Brief Title: Two Different Dietary Approaches in Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Emel Aydan Oral, Instructor, Baskent University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Nutrition
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Time Restricted Feeding; Obesity
Keywords: Obesity; Time restricted feeding; Hormone; Anthropometric measurements
MeSH Terms: conditions — Intermittent Fasting; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Feeding (TRF) (Experimental): Time-restricted feeding program from sunrise to sunset
  Interventions: Behavioral: Time-Restricted Feeding; Behavioral: Extended-Time Feeding
- Extended-Time Feeding (ETF) (Active Comparator): Extended-time feeding program that allows them to eat at any time of the day
  Interventions: Behavioral: Time-Restricted Feeding; Behavioral: Extended-Time Feeding

INTERVENTIONS:
Behavioral: Time-Restricted Feeding — Time-restricted feeding (TRF) is a dietary approach that includes a fasting protocol and a fasting period ranging from 3 to 21 hours during the day . Since there is no standard definition of TRF, fasting/feeding periods vary. In this study, 12-hour fasting and 12-hour feeding period defined by Pureza et al.(11) were taken as the TRF model. In the first 4-week arm of the study, applied a time-restricted feeding program from sunrise to sunset. The daily energy requirements of the participants were calculated individually to lose 5% of their initial weight and the distributions of macronutrients were 45-60% of total energy from carbohydrates, 10-20% as protein and less than 35% from fat.
Behavioral: Extended-Time Feeding — Extended-time feeding program was suggested that allows them to eat at any time of the day. During dietary interventions, a weight loss diet was applied to the participants. The daily energy requirements of the participants were calculated individually to lose 5% of their initial weight and the distributions of macronutrients were 45-60% of total energy from carbohydrates, 10-20% as protein and less than 35% from fat.

SUMMARY:
Objective: In this study, it was aimed to determine the effect of time-restricted feeding on anthropometric measurements and leptin, ghrelin, adiponectin, insulin and cortisol hormone levels in obese women.

Material and Methods: This study was carried out with women who voluntarily accepted to participate in the study who applied to the Baskent University Ankara Hospital Endocrinonogy Outpatient Clinic between September 2019 and October 2020. Women between the ages of 20 and 50, with a body mass index of 29-35 kg/m2, without any chronic disease, who did not have a weight loss diet in the last 6 months, and who had regular night sleep were included in the study. This study was planned as a randomized cross-over design for a total of 9 weeks. Two different dietary interventions, "time-restricted feeding" and "extended-time feeding", were applied to 4 weeks for each group and a week for wash-out period. Anthropometric measurements and hormone levels of individuals were evaluated at the beginning and end of the study.

DETAILED DESCRIPTION:
This study was conducted on volunteers who applied to Başkent University Ankara Hospital Endocrinonogy Outpatient Clinic between September 2019 and October 2020. The study was conducted on women between the ages of 20-50 years, with a body mass index (BMI) between 29-35 kg/m2, sedentary lifestyle, working day shift, regular night sleep habits (bedtime 10:00-12.00 pm; waking time 06:00-08:00 am), without any chronic disease, no dieting history in the last 6 months. Women who were in menopause, with eating disorders, psychiatric illnesses, metabolic and chronic diseases were excluded in the study. As the cross over design study was planned which in the comparison of any quantitative measurement, it was found appropriate to work with at least 29 people in order to reveal a medium to large effect size with a 5% Type I error probability and 86% power probability within the knowledge of the literature. PASS Power Software 3.1.3 for power analysis software was used.A total of 30 women participated in the study. The individuals were randomly divided into 2 groups as Group I (n:15) and Group II (n:15). This study was planned to be a randomized study with a cross-over design for a total of 9 weeks. The study was a two-armed study and two different dietary interventions were applied to the groups: "Time-Restricted Feeding (TRF)" and "Extended-Time Feeding (ETF)". A 1-week washout period was given between two 4-week dietary intervention periods. Ten subjects withdrawn from the study after the first dietary interventon period. A total of 20 people completed the study .At the beginning of the study, a questionnaire (demographic characteristics, educational status, occupation, family history, eating habits and sleep patterns, etc.) was applied to all individuals participating in the study by face-to-face interview method.Since there is no standard definition of TRF, fasting/feeding periods vary. In this study, 12-hour fasting and 12-hour feeding period defined by Pureza et al. were taken as the TRF model. In the first 4-week arm of the study, Group I applied a time-restricted feeding program from sunrise to sunset; for Group II, an extended-time feeding program was suggested that allows them to eat at any time of the day. During dietary interventions, a weight loss diet was applied to the participants. The daily energy requirements of the participants were calculated individually to lose 5% of their initial weight and the distributions of macronutrients were 45-60% of total energy from carbohydrates, 10-20% as protein and less than 35% from fat. Before dietary interventions a 60-minute informative meeting was held by the researcher dietitian, in which the food portion and amount were explained by using the visual food catalog.Anthropometric measurement and body composition were assessed at the beginning and end of each intervention.Serum hormone levels were analyzed at Baskent University Ankara Hospital Biochemistry Laboratory. Blood samples were taken from the patients at the beginning of the study and at the end of each period.Qualitative variables are given as number (S) and percentage (%). Continuous variables (quantitative variables) obtained by measurement are given with mean and standard deviation (¬x̄ ±SD) values. The conformity of the data obtained from the measured quantitative variables to the normal distribution was evaluated with the "Shapiro Wilk Test". Chi-Square (Chi-Square) test was used to determine the relationship or difference between qualitative variables. At the beginning of the study, the "Independent Samples T Test" was used to compare the averages of some quantitative variables according to the diet. "Paired Samples T-Test (T-Test in Dependent Groups)" was used to evaluate the groups within themselves. The criterion of "effect size (d=effect size) obtained from the comparison of dependent/independent groups" was used to determine the degree of effect of dietary interventions on individuals' hormone levels and anthropometric measurements. "Pearson Correlation Coefficent" and "Partial Correlation Coefficent" after removing the initial body weight were used to determine the relationship between quantitative variables. P<0.05 was accepted as the level of significance in all statistical analyses. The data obtained according to the results of the study were evaluated with the SPSS 25 (Statistical Package for Social Sciences) statistical package program.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 20-50 years
* Body mass index (BMI) between 29-35 kg/m2
* Sedentary lifestyle
* Working day shift
* Regular night sleep habits (bedtime 10:00-12.00 pm; waking time 06:00-08:00 am)
* Without any chronic disease
* No dieting history in the last 6 months

Exclusion Criteria:

* Women who were in menopause
* Having eating disorders
* Having psychiatric illnesses
* Having metabolic and chronic diseases

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Leptin | At the beginning and end of each intervention
  ng/mL
Ghrelin | At the beginning and end of each intervention
  pg/mL
Body Weight | At the beginning and end of each intervention
  kg
Body Mass Index (BMI) | At the beginning and end of each intervention
  kg/m2
Body Fat Mass | At the beginning and end of each intervention
  kg

CONTACTS AND LOCATIONS:
Overall Officials: Emel Aydan Oral, Instructor, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravussin E, Beyl RA, Poggiogalle E, Hsia DS, Peterson CM. Early Time-Restricted Feeding Reduces Appetite and Increases Fat Oxidation But Does Not Affect Energy Expenditure in Humans. Obesity (Silver Spring). 2019 Aug;27(8):1244-1254. doi: 10.1002/oby.22518. PMID 31339000
- [Result] de Oliveira Maranhao Pureza IR, da Silva Junior AE, Silva Praxedes DR, Lessa Vasconcelos LG, de Lima Macena M, Vieira de Melo IS, de Menezes Toledo Florencio TM, Bueno NB. Effects of time-restricted feeding on body weight, body composition and vital signs in low-income women with obesity: A 12-month randomized clinical trial. Clin Nutr. 2021 Mar;40(3):759-766. doi: 10.1016/j.clnu.2020.06.036. Epub 2020 Jul 14. PMID 32713721
- [Result] Rynders CA, Thomas EA, Zaman A, Pan Z, Catenacci VA, Melanson EL. Effectiveness of Intermittent Fasting and Time-Restricted Feeding Compared to Continuous Energy Restriction for Weight Loss. Nutrients. 2019 Oct 14;11(10):2442. doi: 10.3390/nu11102442. PMID 31614992
- [Result] Schroder JD, Falqueto H, Manica A, Zanini D, de Oliveira T, de Sa CA, Cardoso AM, Manfredi LH. Effects of time-restricted feeding in weight loss, metabolic syndrome and cardiovascular risk in obese women. J Transl Med. 2021 Jan 6;19(1):3. doi: 10.1186/s12967-020-02687-0. PMID 33407612
- [Result] Stratton MT, Tinsley GM, Alesi MG, Hester GM, Olmos AA, Serafini PR, Modjeski AS, Mangine GT, King K, Savage SN, Webb AT, VanDusseldorp TA. Four Weeks of Time-Restricted Feeding Combined with Resistance Training Does Not Differentially Influence Measures of Body Composition, Muscle Performance, Resting Energy Expenditure, and Blood Biomarkers. Nutrients. 2020 Apr 17;12(4):1126. doi: 10.3390/nu12041126. PMID 32316561
- [Result] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952